CLINICAL TRIAL: NCT04259463
Title: The Influence of Sedation and General Anesthesia to Patients' Psycho-emotional State Undergoing Wisdom Teeth Extraction
Status: Completed | Type: Observational
Sponsor: Inesa Astramskaitė (Other)
Responsible Party: Sponsor-Investigator, Inesa Astramskaitė, DDS Inesa Astramskaite Januseviciene, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: BEC-OF-03
Record Dates: First submitted 2020-01-30; First posted 2020-02-06 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Teeth, Impacted; Tooth-loss; Anxiety; Fear
MeSH Terms: conditions — Tooth, Impacted; Anodontia; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Concious sedation: Patients undergoing third molars extraction under concious sedation. The patient is fully familiarized with the sedation procedure. The anesthesiologist suppresses the patient's consciousness with the help of intravenous medication;
  Interventions: Procedure: Third molars extraction
- Full anesthesia: Patients undergoing third molars extraction under full anesthesia. . The patient is fully acquainted with the procedure of general anesthesia. It is a controlled state of unconsciousness when protective reflexes disappear, the patient cannot breathe and does not respond to verbal commands. A special intubation tube is introduced into the airways.
  Interventions: Procedure: Third molars extraction

INTERVENTIONS:
Procedure: Third molars extraction — Third molars extractions with concious sedation or general anesthesia

SUMMARY:
The aim of the study is to evaluate, wheather the sedation or general anesthesia in third molar extractions influence the patient's psycho-emotional status. It is believed that the type of anesthesia may influence not only the psycho-emotional status after the procedure, but also before the procedure.

DETAILED DESCRIPTION:
A prospective pilot study was conducted on adult patients who were admitted to the Faculty of Surgery at LSMU KK hospital for removal of all four wisdom teeth with sedation or general anesthesia. The patients were given one day to complete the given questionnaires. They were asked to complete three questionnaires: a) before the surgery, i.e. at the time the patient was hospitalized; b) the same day prior to surgery; c) ten days after the surgery. The operating doctor also filled out a questionnaire ten days after the surgery.

The aim of the study is to evaluate, wheather the sedation or general anesthesia in third molar extractions influence the patient's psycho-emotional status. It is believed that the type of anesthesia may influence not only the psycho-emotional status after the procedure, but also before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years;
* Indicated removal of all 4 wisdom teeth;
* Non-use of NSAIDs, anticoagulants;
* No acute inflammation in the operated area;
* No history of common conditions that contraindicate oral surgery. For example, uncontrolled diabetes, cardiovascular disease;
* Patients agreed to participate in the study.

Exclusion Criteria:

* Pregnant, breastfeeding women;
* Individuals, formerly treated with radiation;
* Patients who participated in studies related to the assessment of psycho-emotional status;
* Patients with obvious mental, intellectual or physical disabilities limiting the participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients, undergoing the third molars extraction with sedation or general anesthesia, that meet the inclusion criteria are randomly selected.
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Anesthesia effect on patients pre-operative psycho-emotional status: questionnaire | baseline, pre-intervention/procedure/surgery
  Anesthesia effect on patients pre-operative psycho-emotional status. The following scales are used: Universal Scale in Oral Surgery for psycho-emotional rating (1-3 raiting with higher rating meaning more negative psycho-emotional status); Modified Corah's Dental Anxiety Questionnaire (1-5 scores with with higher rating meaning more negative psycho-emotional status); visual analogue scales on fear of tooth extraction and fear of general anesthesia (1-5 scores with higher rating meaning higher fear)
Anesthesia effect on patients pre-operative psycho-emotional status: questionnaire | immediately after the intervention/procedure/surgery
  Anesthesia effect on patients pre-operative psycho-emotional status. The following scales are used: Universal Scale in Oral Surgery for psycho-emotional rating (1-3 raiting with higher rating meaning more negative psycho-emotional status); Modified Corah's Dental Anxiety Questionnaire (1-5 scores with with higher rating meaning more negative psycho-emotional status); visual analogue scales on fear of tooth extraction and fear of general anesthesia (1-5 scores with higher rating meaning higher fear)
Anesthesia effect on patients post-operative psycho-emotional status: questionnaire | 10 days after after the intervention/procedure/surgery
  Anesthesia effect on patients post-operative psycho-emotional status. The following scales are used: Universal Scale in Oral Surgery for psycho-emotional rating (1-3 raiting with higher rating meaning more negative psycho-emotional status); Modified Corah's Dental Anxiety Questionnaire (1-5 scores with with higher rating meaning more negative psycho-emotional status); visual analogue scales on fear of tooth extraction and fear of general anesthesia (1-5 scores with higher rating meaning higher fear). Also the pain that was felt immediately after the procedure, 6 hours after the procedure, 24 hours after the procedure, 2-10 days after the procedure was evaluated. The linear scale of 10cm was used, where the less points ment lower pain. Patient had to point the vertical dash on a line to represent the pain

CONTACTS AND LOCATIONS:
Overall Officials: Inesa Astramskaite Januseviciene, DDS, Study Director — LUHS
Locations (1):
- Maxillofacial Surgery, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No